CLINICAL TRIAL: NCT00812279
Title: A Controlled, Randomised, Open-label, 3-arm Parallel Single-centre Confinement Study to Investigate Exposure to Selected Smoke Constituents in Smokers Switching From Conventional Cigarettes to SMAR Cigarettes for 5 Days
Brief Title: Investigate the Exposure to Selected Smoke Constituents in Smokers Switching to Distillation Based Smoking Article
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: YVD-CS01-EU
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Smoking
Keywords: Smokers with acceptable health conditions
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. SMAR (Experimental): Subjects will be allowed to smoke SMAR without any limit on consumption during the designated smoking times.
  Interventions: Other: Distillation based smoking article (SMAR cigarette)
- 2 Conventional cigarette (CC) (Active Comparator): Subjects will be allowed to smoke without any limit on consumption during the designated smoking times.
  Interventions: Other: conventional cigarette
- 3. smoking cessation (SC) (Active Comparator): Subjects will not be allowed to smoke any cigarettes or to use any other nicotine/tobacco-containing products during the 5 days following randomisation.
  Interventions: Other: smoking cessation

INTERVENTIONS:
Other: Distillation based smoking article (SMAR cigarette) — Subjects randomised to the SMAR arm will be trained by the site staff on the usage of SMAR and the corresponding lighter prior to smoking the first SMAR. Subjects will be allowed to smoke SMAR without any limit on consumption during the designated smoking times but have to request each SMAR from the site staff when they wish to smoke.
  Arms: 1. SMAR
Other: conventional cigarette — Subjects randomised to the CC arm will continue to smoke their preferred CC brand during the exposure period. Subjects will be allowed to smoke without any limit on consumption during the designated smoking times but will have to request each CC from the site staff when they wish to smoke.
  Arms: 2 Conventional cigarette (CC)
Other: smoking cessation — Subjects will not be allowed to smoke any cigarettes or to use any other nicotine/tobacco-containing products during the 5 days following randomisation.
  Arms: 3. smoking cessation (SC)

SUMMARY:
The overall purpose of this clinical study conducted in confinement under well-defined conditions is to obtain initial data on the levels of human body exposure to selected smoked constituents of the SMAR cigarette.

The main objective of this study is to compare the biomarkers of exposure to cigarette smoke constituents in smokers switching to SMAR and to biomarkers in smokers of conventional cigarettes (CC). The biomarkers of exposure will be measured in blood and urine samples collected from the subjects. Moreover, the biomarkers in subjects smoking conventional or SMAR cigarettes will be compared with those biomarkers in smokers who stop smoking for 5 days. The short term safety of this new product will also be evaluated.

DETAILED DESCRIPTION:
This is a controlled, randomised, open-label, 3-arm parallel single centre confinement study to investigate exposure to selected smoke constituents in smokers switching from CC to SMAR for 5 days.

112 eligible subjects will be randomised to the 3 study arms: SMAR, conventional cigarettes (CC) and smoking cessation (SC) in a 2:1:1 ratio.

Following the screening visit (within 4 weeks prior to the day of admission), the study will be run over an 8-day period in a confined environment, consisting of the admission day (D-2), a 2-day baseline period (D-1 and D0), and a 5-day exposure period (D1 to D5). Subjects will be discharged in the morning of D6. From the discharge of the subject, a 7-day safety follow-up period will be carried out (until D13).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian adult smokers (male and female), with acceptable health conditions, aged from 23 to 55 years who usually smoke 10 to 30 non-mentholated conventional cigarettes (with a maximum ISO tar yield of 10 mg) per day, for at least the last 5 consecutive years, will be enrolled in this study.

Exclusion Criteria:

* women of childbearing potential must be excluded if:Subject is pregnant (does not have negative pregnancy tests at screening and at D-2) or breastfeeding/ subject does not agree to use an acceptable method of effective contraception: intrauterine device, intrauterine system, established use of oral/injectable/implantable/ transdermal hormonal methods, barrier methods of contraception (condoms, occlusive caps) with spermicidal foam/gel/film/suppository, vasectomised partner or true abstinence (periodic abstinence and withdrawal are not effective methods) until the end of the safety follow-up period.

Ages: 23 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To demonstrate a reduction in the three primary biomarkers of exposure: Carboxyhaemoglobin concentration in blood, Urinary excretion of S-phenylmercapturic acid and urinary excretion of NNAL and NNAL-glucuronides (total NNAL) | 5 days

SECONDARY OUTCOMES:
To explore changes from baseline COHb, S-PMA, and total NNAL in the three study arms in the course of the study | 5 days
To explore changes from baseline in the three study arms with regard to urinary excretion of biomarkers of exposure to several other smoke constituents. | 5 days
To assess urinary excretion of nicotine and its five major nicotine metabolites in the three study arms | 5 days
To assess nicotine and cotinine concentrations in plasma in the three study arms To compare levels of all biomarkers of exposure in the SMAR arm to those in the smoking cessation (SC) arm | 5 days
To assess the mutagenicity potential in urine at the end of the study in the three study arms | 5 days
To monitor blood pressure, pulse rate, electrocardiogram, clinical laboratory parameters (standard clinical biochemistry, standard haematology and urine analysis), and adverse events | 5 days
To investigate craving and withdrawal symptoms as well as pulmonary symptoms in all three study arms by means of questionnaires | 5 days
To investigate change in cytochrome P450 1A2 (CYP1A2) activity from D0 to D5 in the three study arms | 5 days
To assess and compare human smoking topography (HST) in smokers before and after switching to SMAR | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Jarus-Dziedzic, MD, Principal Investigator — MTZ Clinical Research Inc (Warsaw, Poland)
Locations (1):
- MTZ Clinical Research Inc., Warsaw, Poland

REFERENCES:
- [Result] Ludicke F, Haziza C, Weitkunat R, Magnette J. Evaluation of Biomarkers of Exposure in Smokers Switching to a Carbon-Heated Tobacco Product: A Controlled, Randomized, Open-Label 5-Day Exposure Study. Nicotine Tob Res. 2016 Jul;18(7):1606-13. doi: 10.1093/ntr/ntw022. Epub 2016 Jan 27. PMID 26817490